CLINICAL TRIAL: NCT01698333
Title: An Open Label Evaluation of the Adrenal Suppression Potential and Pharmacokinetic Properties of Twice Daily 122-0551 in Subjects With Plaque Psoriasis Receiving Two Weeks of Treatment
Brief Title: Pharmacokinetics of 122-0551 and Its Effects on Adrenal Suppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122-0551-202
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Plaque Psoriasis
Keywords: 122-0551; steroid; HPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 122-0551 (Experimental)
  Interventions: Drug: 122-0551

INTERVENTIONS:
Drug: 122-0551 — Applied twice daily for 2 weeks

SUMMARY:
Adrenal suppression effects of corticosteroids are among the most important safety concerns for this group of products. This study is designed to determine the adrenal effects of the investigational formulation of 122-0551 and characterize the steady state pharmacokinetics of the formulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of stable plaque psoriasis

Exclusion Criteria:

* Subject has spontaneously improving or rapidly deteriorating plaque psoriasis
* Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis
* Subject has used any phototherapy, photo-chemotherapy or systemic psoriasis therapy within 30 days prior to initiation of treatment
* Subject has used systemic corticosteroids or topical, inhaled, intranasal corticosteroids within 30 days and 14 days, respectively, prior to study screening
* Subject has had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to initiation of treatment
* Subject has used topical psoriatic therapy including tar, anthralin, retinoids, vitamin D analogs (e.g., Dovonex®) within 14 days prior to initiation of treatment
* Subject has used emollients/moisturizers on areas to be treated within one day prior to initiation of treatment
* Subject is currently using lithium or Plaquenil (hydroxychloroquine)
* Subject is currently using a beta-blocking medication (e.g., propranolol) or angiotensin converting enzyme (ACE) inhibitors (e.g., lisinopril) at a dose that has not been stabilized
* Subject is pregnant, nursing or planning a pregnancy during the study period
* Subject is currently enrolled in an investigational drug, biologic or device study
* Subject has received an investigational drug, biologic or an investigational device within 30 days prior to study start
* Subject has been previously enrolled in this study and treated with the test article
* Subject has an irregular sleep schedule or works night shifts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syd Dromgoole, PhD, Study Director — Therapeutics, Inc.
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - Therapeutics Clinical Research, San Diego, California
  - DermResearch, Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: April 2012 to March 2013
  The location of clinical sites included private dermatology clinics and clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were enrolled into the study.
Period: Overall Study
Arm/Group | 122-0551
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) population included all participants enrolled in the study who were dispensed and applied test article at least once and had at least one follow-up visit after the Baseline visit (Visit 2). All 25 enrolled subjects were included in the ITT population.
Arm/Group | 122-0551
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 21
  Race: Asian | 3
  Race: Islander | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Hypothalamic-Pituitary-Adrenal (HPA) Axis Response
Description: HPA axis response to stimulation by cosyntropin, dichotomized to "normal" and "abnormal". Laboratory evidence of abnormal HPA axis response is defined as a 30-minute post-stimulation serum cortisol level that is ≤ 18 μg/dL at the end of study.
Time Frame: Day 15
Population: Analysis shown is based on the ITT population, defined as all enrolled participants who applied at least one dose of the test article and returned for at least one post-Baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | 122-0551
Number analyzed (Participants) | 25
Participants
  Normal | 19
  Abnormal | 6

ADVERSE EVENTS:
Time Frame: AEs were collected from study screening (performed 20 days or more prior to baseline/first dose) to end of study treatment or participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The Safety population included all subjects enrolled in the study who were dispensed the test article at least once. Each subject counted once for each AE Term.
Arm/Group | 122-0551
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 8/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 122-0551 (N=25)
Pharyngitis (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1)
ACTH Stimulation Test Abnormal (Investigations) | 6 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 30 days prior to public dissemination. The PI may not disclose previously undisclosed confidential information other than study results.